CLINICAL TRIAL: NCT06150209
Title: A Controlled Data Collection and Prospective Treatment Study to Evaluate the Efficacy of Vendaje in the Management of Foot Ulcers in Diabetic Patients.
Brief Title: A Controlled Prospective Treatment Study to Evaluate the Efficacy of Vendaje.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioStem Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Diabetic Foot Ulcer/1
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Time points to wound closure compared to retrospective standard of care closure times. If closure is not achieved the reduction in wound volume will be evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Vendaje (Other): application of Vendaje
  Interventions: Device: Vendaje

INTERVENTIONS:
Device: Vendaje — Dehydrated Human Amniotic Membrane

SUMMARY:
The Goal of this study is to evaluate the wound volume reduction rate and the time to closure when using Vendaje to manage diabetic wounds.

The participants will be treated weekly for up to 12 weeks.

The data will be compared to retrospective Standard of care data from similarly controlled studies

DETAILED DESCRIPTION:
Patients will be recruited by the site PIs and will be educated on the details of the study through the use of a detailed And IRB approved informed consent.

They must meet the inclusion/exclusion criteria which includes appropriate testing for perfusion and control of diabetes.

Once accepted a screening visit without Vendaje treatment but SOC treatment to determine if closure with SOC will be adequate.

If the SOC screen fails a threat protocol begins for up to 12 weeks or closure.

data will be collected using digital planimetry and also recorded in a research binder with CRFs provided.

A final visit 2 weeks after closure or end of 12 weeks will provided information related to wound recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Have adequate vascular perfusion to the surgical site limb as defined by one of the following in order of preference.

   1. Ankle Brachial Pressure Index (ABI) > 0.65 < 1.3.
   2. Toe Pressure of greater than 40mmHg.
   3. TcPO2 of greater than 40mmGg.
3. Skin Perfusion Pressure (SPP) > 30. (Calculations will be made using measurements from both dorsalis pedis arteries and posterior tibial arteries of affected limbs).
4. Presence of a diabetic foot ulcer extending through the full thickness of the skin but not down to muscle, tendon or bone. The largest ulcer will be designated the index ulcer and the only one included in the study. If other ulcerations are present on the same leg they have to be more than 2 cm apart from the index ulcer.
5. Study ulcer (i.e. current episode of ulceration) has been present for at least one month prior to the initial screening visit, and is excluded if it has undergone 1 month of continuous high strength offloading therapy over its duration..
6. Study ulcer is a minimum of 1 cm2 and a maximum of 25 cm2 at the application visit.
7. The target ulcer has been treated with standard of care and offloading therapy for at least 14 days prior to application.
8. Ulcer has a clean, granulating base with minimal adherent slough at the randomization visit.
9. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
10. Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
11. Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Study ulcer exhibits clinical signs and symptoms of infection.
3. Study ulcer, in the opinion of the investigator, is suspicious for cancer should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
4. Patients with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
5. Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding Screening. (All Covid-19 Vaccines are exempt as investigational drugs under this protocol)
6. History of radiation at the ulcer site.
7. Study ulcer has been previously treated with tissue engineered materials (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days
8. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
9. Patients who are unable to understand the aims and objectives of the trial.
10. The presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
11. Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus are excluded.
12. Pregnant or breast feeding.
13. Currently taking medications which could affect graft incorporation. (supervising physicians' discretion)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Time Closure in Diabetic foot ulcers Managed with Vendaje | 12 weeks of treatment
  The effect on closure rates of diabetic foot ulcers when Vendaje is applied to the wound bed

SECONDARY OUTCOMES:
Reduction of wound volume in diabetic foot ulcers treated with Vendaje | 12 weeks of treatment
  Effect of Venaje on the volume reduction of diabetic foot ulcers when Vendaje is applied.

CONTACTS AND LOCATIONS:
Overall Officials: John Starinski, DPM, Principal Investigator — BioStem Technologies

IPD SHARING:
Plan to Share IPD: No
Data will be processed and published.